CLINICAL TRIAL: NCT03631524
Title: Using Telerehabilitation Tools to Deliver Quality Therapy to Patients Under Infective Isolation Precautions
Acronym: IsoRehab2018
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Geoffrey Sithamparapillai Samuel, Consultant, Department of Rehabilitation Medicine, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/2994
Record Dates: First submitted 2018-08-03; First posted 2018-08-15 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Deconditioning, Isolation Precautions
Keywords: deconditioning, isolation precautions, telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Two arm single blinded RCT
Who Masked: Outcomes Assessor
Masking Description: Block Randomisation, Initial and final outcome assessors blinded to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (No Intervention): The control arm will be subject to the same assessments as the treatment arm at the start and end of the two week period. They will receive standard care in the ward including physiotherapy as prescribed by the managing team
- Intervention arm (Experimental): The treatment arm will be given up to 1 hour of physiotherapist-prescribed resistive training exercises administered via a telerehabilitation device per day in addition to standard therapy for a total of 10 sessions over a 2 week period. They will be evaluated for motor strength, activity of daily living performance, mood and perceived level of health.
  Interventions: Device: Telerehabilitation

INTERVENTIONS:
Device: Telerehabilitation — The treatment arm will be given up to 1 hour of physiotherapist-prescribed resistive training exercises administered via a telerehabilitation device per day in addition to standard therapy for a total of 10 sessions over a 2 week period.
  Arms: Intervention arm

SUMMARY:
Single blinded Randomised Controlled trial comparing standard therapy to the intervention of up to 1 hour of physiotherapist-prescribed resistive training exercises administered via a telerehabilitation device per day in addition to standard therapy for a total of 10 sessions over a 2 week period. Total recruitment: 60 patients.

DETAILED DESCRIPTION:
This is a single blinded randomised control trial. From August 2018 to March 2019, a total of 60 subjects, who match the inclusion exclusion criteria, will be recruited from patients transferred to the SGH Isolation wards.

They will be randomly assigned to control or treatment arm based on a block randomisation strategy predetermined and held by an independent party.

The treatment arm will be given up to 1 hour of physiotherapist-prescribed resistive training exercises administered via a telerehabilitation device per day in addition to standard therapy for a total of 10 sessions over a 2 week period. They will be evaluated for motor strength, activity of daily living performance, mood and perceived level of health.

The control arm will be subject to the same assessments as the treatment arm at the start and end of the two week period. They will receive standard care in the ward including physiotherapy as prescribed by the managing team.

The assessors will be blinded to the arm of the study the subjects will be assigned to and will be independent of the terating physiotherapist.

1.1. Hypothesis We propose that for patients with deconditioning after a prolonged period of hospitalization and needing inpatient isolation precautions, that a 2-week course of daily, up to 1-hour long, physiotherapist-developed resistive training exercises will result in a 20% improvement in the motor power and a corresponding improvement in motor functioning and the perceived quality of life compared to a control group receiving standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Able to give consent

  * Admitted to hospital for at least 5 days
  * MMT power grading 2-4/5
  * Isolated for prevention of transmission of MDROs

Exclusion Criteria:

* • Unable or unwilling to consent for the trial

  * Assessed by managing team to be fit for discharge within the next 2 weeks
  * Pregnant women
  * Underlying medical disorders that result in pre-existing lower limb weakness

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Manual motor power testing | 2 weeks
  To assess change in the motor function level (as determined by
  1. Medical Research Council (MRC) Manual Muscle Testing (MMT)) at the end of 2 weeks of assessment.
  2. To assess change of quadriceps strength using a handheld dynamometer at the end of 2 weeks of assessment

SECONDARY OUTCOMES:
Volume of therapy | 2 weeks
  The number of repetitions of each exercise will be used as corraborative evidence of progress during therapy.
Functional Independence Measure | 2 weeks
  The FIM Provides a uniform system of measurement for disability based on the International Classification of Impairment, Disabilities and Handicaps; measures the level of a patient's disability and indicates how much assistance is required for the individual to carry out activities of daily living based on their score in 18 categories (13 motor and 5 cognitive function items). Each category or item is rated on a 7-point scale (1 = total assistance required, 7 = fully independent).
  Coster, W. J., Haley, S. M., et al. (2006). "Measuring patient-reported outcomes after discharge from inpatient rehabilitation settings." J Rehabil Med 38(4): 237-242.
Level of anxiety/ depression | 2 weeks
  Hospital Anxiety and Depression Score. The HADS is a fourteen item clinical assessment scale to assess levels of anxiety and depression. Seven of the items relate to anxiety and seven relate to depression.
  Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses an ordinal scale.
  A number of researchers have explored HADS data to establish the cut-off points for diagnosis of anxiety or depression. A systematic review of a large number of studies identified a cut-off point of 8/21 for anxiety or depression. For anxiety (HADS-A) this gave a specificity of 0.78 and a sensitivity of 0.9. For depression (HADS-D) this gave a specificity of 0.79 and a sensitivity of 0.83.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey S Samuel, MBBS, Principal Investigator — Singhealth Pte Ltd

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morgan DJ, Diekema DJ, Sepkowitz K, Perencevich EN. Adverse outcomes associated with Contact Precautions: a review of the literature. Am J Infect Control. 2009 Mar;37(2):85-93. doi: 10.1016/j.ajic.2008.04.257. PMID 19249637
- [Background] Ploutz-Snyder LL, Downs M, Ryder J, Hackney K, Scott J, Buxton R, Goetchius E, Crowell B. Integrated resistance and aerobic exercise protects fitness during bed rest. Med Sci Sports Exerc. 2014 Feb;46(2):358-68. doi: 10.1249/MSS.0b013e3182a62f85. PMID 24441215